CLINICAL TRIAL: NCT00770185
Title: A Phase II Study of Ridaforolimus in Patients With Metastatic And/Or Locally Advanced Recurrent Endometrial Cancer
Brief Title: Ridaforolimus in Treating Patients With Recurrent Metastatic and/or Locally Advanced Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I192; CAN-NCIC-IND192 (Registry Identifier: NCI US - Physician Data Query); ARIAD-CAN-NCIC-IND192 (Other: Ariad); CDR0000614597 (Other: PDQ)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Endometrial Cancer
Keywords: endometrial adenocarcinoma; endometrial adenosquamous cell carcinoma; endometrial clear cell carcinoma; endometrial papillary carcinoma; recurrent endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — ridaforolimus; Gene Expression Profiling; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ridaforolimus (Experimental): oral ridaforolimus 40 mg days 1-5 each week (once daily for 5 consecutive days every week; cycle arbitrarily defined as a 4 week period)
  Interventions: Drug: ridaforolimus; Genetic: gene expression analysis; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: ridaforolimus — oral ridaforolimus 40 mg days 1-5 each week (once daily for 5 consecutive days every week; cycle arbitrarily defined as a 4 week period)
Genetic: gene expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Ridaforolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying the side effects of ridaforolimus and to see how well it works in treating patients with recurrent metastatic and/or locally advanced endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the efficacy, in terms of objective response rate, of ridaforolimus, in patients with recurrent metastatic and/or locally advanced endometrial cancer.
* To assess the adverse events, time to progression, and response duration of this drug in these patients.
* To correlate objective tumor response with PTEN expression and other potential markers in primary tumor tissue from these patients.

OUTLINE: This is a multicenter study.

Patients receive oral ridaforolimus once daily on days 1-5 for 4 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Archived tumor tissue samples (paraffin block or unstained slides) are analyzed for PTEN gene expression and other mTOR pathway elements to explore possible markers of response or non-progression by immunohistochemistry.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed endometrial cancer, including any 1 of the following subtypes:

  * Adenocarcinoma

    * Papillary serous
    * Papillary
    * Villoglandular
    * Mucinous
    * Clear cell
  * Endometrioid
  * Adenosquamous carcinoma
* Recurrent or metastatic and/or locally advanced disease
* Incurable disease by standard therapies
* Clinically and/or radiologically documented disease within the past 28 days (35 days if negative), defined as ≥ 1 unidimensionally measurable disease site meeting 1 of the following criteria:

  * At least 20 mm by x-ray or physical exam
  * At least 10 mm by spiral CT scan
  * At least 20 mm by non-spiral CT scan
* Available tumor tissue (paraffin block or unstained slides) from primary tumor
* No uterine sarcoma (leiomyosarcoma), mixed müllerian tumor (MMT), and/or adenosarcoma
* No known brain metastases

  * Clinical suspicion of CNS involvement requires a head CT scan

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN
* Creatinine ≤ 1.25 times ULN OR creatinine clearance ≥ 50 mL/min
* Fasting serum cholesterol ≤ 9.0 mmol/L
* Fasting triglycerides ≤ 4.56 mmol/L
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Accessible for treatment and follow up (e.g., 1 ½ hours driving distance from participating center)
* No upper gastrointestinal or other condition that would impair swallowing or absorption of oral medication
* No serious illness or medical condition that would not permit the patient to be managed according to the protocol, including, but not limited to, any of the following:

  * History of significant neurologic or psychiatric disorder (e.g., uncontrolled psychotic disorders) that would impair the ability to obtain consent or limit compliance with study requirements
  * Active uncontrolled or serious infection
  * Active peptic ulcer disease
  * Myocardial infarction within the past 6 months, congestive heart failure (even if medically controlled), unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, or uncontrolled hypertension
  * Pulmonary disease requiring oxygen
  * HIV infection or other immune deficiency
  * Other medical conditions that might be aggravated by study treatment
* No history of other malignancies, except adequately treated nonmelanoma skin cancer, curatively treated carcinoma in situ of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years
* No known hypersensitivity to the study drug or its components

PRIOR CONCURRENT THERAPY:

* At least 7 days since prior hormonal therapy (progestational or aromatase inhibitor) as either adjuvant therapy or for treatment of metastatic disease
* At least 21 days since prior major surgery and recovered
* At least 28 days since prior radiotherapy and recovered

  * Prior low-dose palliative radiotherapy allowed
* At least 4 months since prior adjuvant chemotherapy
* No prior mTOR inhibitors
* No prior or concurrent chemotherapy for metastatic or recurrent disease
* More than 7 days since prior and no concurrent CYP3A4 inhibitors including, but not limited to, any of the following:

  * Azole antifungals (i.e., ketoconazole, itraconazole, miconazole, fluconazole)
  * HIV protease inhibitors (i.e., indinavir, saquinavir, ritonavir, atazanavir, nelfinavir)
  * Clarithromycin
  * Verapamil
  * Erythromycin
  * Delavirdine
  * Diltiazem
  * Nefazodone
  * Telithromycin
* More than 12 days since prior and no concurrent CYP3A4 inducers including, but not limited to, any of the following:

  * Rifampin
  * Phenytoin
  * Rifabutin
  * St. John's wort
  * Carbamazepine
  * Efavirenz
  * Phenobarbital
  * Tipranavir
* At least 14 days since prior and no concurrent investigational drugs or anticancer therapy (e.g., immunotherapy, biological response modifiers [excluding hematopoietic growth factors], and systemic hormonal therapy)
* No concurrent CYP3A4 substrates

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-11-13 (Actual); Primary Completion 2012-03-19 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
Objective response measured by RECIST criteria | every 8 weeks
  After every second cycle
Adverse events | 4 years
  Adverse events will be monitored and assessed from the time of the first dose with overall results being assessed at final analysis.
Time to progression | 4 years
Correlation between objective tumor response with PTEN expression and other potential markers | 4 years
  will be assessed overall at the time of completion of therapy and final analysis.

SECONDARY OUTCOMES:
Response duration | 4 years
  After progression with overall results assessed at final analysis

CONTACTS AND LOCATIONS:
Overall Officials: Amit M. Oza, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (11):
- Canada (11):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tsoref D, Welch S, Lau S, Biagi J, Tonkin K, Martin LA, Ellard S, Ghatage P, Elit L, Mackay HJ, Allo G, Tsao MS, Kamel-Reid S, Eisenhauer EA, Oza AM. Phase II study of oral ridaforolimus in women with recurrent or metastatic endometrial cancer. Gynecol Oncol. 2014 Nov;135(2):184-9. doi: 10.1016/j.ygyno.2014.06.033. Epub 2014 Aug 28. PMID 25173583